CLINICAL TRIAL: NCT02591940
Title: Proof of Concept of Model Based Cardiovascular Prediction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: German Heart Institute (Other)
Collaborators: Bambino Gesù Hospital and Research Institute (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: Cardioproof
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Modeling; Aortic Coarctation; Aortic Valve Disease; Cardiovascular MRI
Keywords: cardiovascular modeling; aortic coarctation; aortic valve disease
MeSH Terms: conditions — Aortic Coarctation; Aortic Valve Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aortic Coarctation: interventional treatment in heart catheter (stenting/angioplasty) surgical repair of coarctation
  Interventions: Procedure: Surgery or Treatment by Heart Catheter
- Aortic Valve Disease: surgical repair in aortic valve disease (reconstruction/valve replacement)
  Interventions: Procedure: Surgery or Treatment by Heart Catheter

INTERVENTIONS:
Procedure: Surgery or Treatment by Heart Catheter

SUMMARY:
CARDIOPROOF is a proof-of-concept project that consolidates the outcomes of previous virtual physiological human (VPH) projects and checks the applicability and effectiveness of available predictive modelling and simulation tools, validating them in interrelated clinical trials conducted in three European centres of excellence in cardiac treatment (from Germany, Italy and the UK). CARDIOPROOF focuses on patients with aortic valve disease and aortic coarctation, which, if left untreated, can ensue irreversible heart failure. As a result treatment becomes mandatory, but optimum timing and the best type of treatment still remain difficult to determine. With more than 50.000 interventions per year within the EU, the diseases addressed by CARDIOPROOF have a significant socio-economic impact. Present clinical guidelines are highly complex and rely mostly on imaging diagnostics and clinical parameters, without benefiting, as yet, from patient-specific disease modelling based prediction. CARDIOPROOF goes beyond the current state of the art by conducting validation trials aimed at covering and comparing the complete spectrum of cardiovascular treatment, predicting the evolution of the disease and the immediate and mid-term outcome of treatment. Operational clustering is going to provide a seamless clinical solution that applies different modeling methods to realize the potential of personalised medicine taking into account user-friendliness as a key component of clinical usability. CARDIOPROOF's goal is to provide first-hand data on comparative cost-effectiveness and clinical efficacy of the most advanced VPH approaches compared to conventional diagnostics and treatment algorithms, thus accelerating the deployment of VPH methods in clinical environments, and bring to maturity holistic patient-specific computer-based predictive models and simulations.

ELIGIBILITY:
Inclusion Criteria:

* patients with the need for surgical or interventional treatment with Aortic Coarctation
* patients with the need for aortic valve disease surgery

  * both according to current treatment guidelines

Exclusion Criteria:

* contraindications for MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the need for surgical or interventional treatment with Aortic Coarctation, as well as patients with the need for aortic valve disease surgery, both according to current treatment guidelines.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Comparative Cost effectiveness between regular treatment vs. simulated alternative treatment | 1 week up to 1 year
Predicted (simulated) vs. real haemodynamic 4D flow profile (treatment outcome) | 1 week up to 1 year

SECONDARY OUTCOMES:
Calculated Vessle comliance | 1 week up to 1 year
Calculated External and Internal Heart Power | 1 week up to 1 year
Number of Participants with Aortic Coarctation with Arterial Hypertension | 1 week up to 1 year

REFERENCES:
- [Derived] Runte K, Brosien K, Schubert C, Nordmeyer J, Kramer P, Schubert S, Berger F, Hennemuth A, Kuehne T, Kelm M, Goubergrits L. Image-Based Computational Model Predicts Dobutamine-Induced Hemodynamic Changes in Patients With Aortic Coarctation. Circ Cardiovasc Imaging. 2021 Feb;14(2):e011523. doi: 10.1161/CIRCIMAGING.120.011523. Epub 2021 Feb 16. PMID 33591212
- [Derived] Nordmeyer S, Hellmeier F, Yevtushenko P, Kelm M, Lee CB, Lehmann D, Kropf S, Berger F, Falk V, Knosalla C, Kuehne T, Goubergrits L. Abnormal aortic flow profiles persist after aortic valve replacement in the majority of patients with aortic valve disease: how model-based personalized therapy planning could improve results. A pilot study approach. Eur J Cardiothorac Surg. 2020 Jan 1;57(1):133-141. doi: 10.1093/ejcts/ezz149. PMID 31131388
- [Derived] Fernandes JF, Goubergrits L, Bruning J, Hellmeier F, Nordmeyer S, da Silva TF, Schubert S, Berger F, Kuehne T, Kelm M; CARDIOPROOF Consortium. Beyond Pressure Gradients: The Effects of Intervention on Heart Power in Aortic Coarctation. PLoS One. 2017 Jan 12;12(1):e0168487. doi: 10.1371/journal.pone.0168487. eCollection 2017. PMID 28081162